CLINICAL TRIAL: NCT03971214
Title: Pilot Study on PD-1 Inhibitors Consolidation After Standard First-line Chemotherapy and Radiotherapy in Extensive-stage Small Cell Lung Cancer
Brief Title: PD-1 Inhibitors Consolidation in Extensive-stage Small Cell Lung Cancer
Acronym: PICARES
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Luhua Wang, Professor, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCC1835
Record Dates: First submitted 2019-05-29; First posted 2019-06-03 (Actual); Last update posted 2019-06-04 (Actual); Status verified 2019-06

CONDITIONS: Extensive-stage Small Cell Lung Cancer; Radiotherapy; Immunotherapy
Keywords: small cell lung cancer; radiotherapy; PD-1 inhibitor
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — Drug Therapy; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PD-1 inhibitor JS-001 consolidation for SCLC (Experimental): The extensive-stage SCLC patients will receive PD-1 inhibitor JS-001 treatment after standard first-line chemotherapy, chest radiotherapy ± SABR for metastasis disease, and propylactic cranial irradiation untill disease progression or death.
  Interventions: Drug: PD-1 inhibitor JS-001

INTERVENTIONS:
Drug: PD-1 inhibitor JS-001 — The extensive-stage SCLC patients will receive PD-1 inhibitor treatment after standard first-line chemotherapy, chest radiotherapy ± SABR for metastasis disease, and propylactic cranial irradiation untill disease progression or death.
  Other Names: chemotherapy; radiotherapy; SABR; propylactic cranial irradiation

SUMMARY:
The prognosis of extensive-stage small cell lung cancer is still very poor, even for those who received platinum-based chemotherapy and chest radiotherapy. 2-year survival rate of these patients is only about 10%. Therefore, this study aims to explore a comprehensive treatments with low toxicity to further improve the efficacy for these paitents with PD-1 inhibitor.

DETAILED DESCRIPTION:
The study is a prospective pilot trial. The purpose of this study is to evaluate the safety and efficacy of PD-1 inhibitor consolidation in extensive-stage small cell lung cancer paitents who received standard first-line chemotherapy and chest radiotherapy ± SABR for metastasis disease.

The primary endpoint is the safety and objective response rate of treatment. The secondary objectives are progression free survival(PFS), overall survial. The exploratory end point includes the correlation of PD-1 expression on the tumor tissue, and the TMB, Immune Repertoire sequencing derived from the tumor tissue and the blood sample with the efficacy of treatent. The plan for collection of tumor tissue and blood at baseline at different stages during or after treatment was defined in the protocol.

The PICCARE-trial has been designed by National Cancer Center/Cancer Hospital, Chinese Academy of Medical Sciences, Peking Union Medical College, and the hypothesis is PD-1 inhibitor consolidation was safe and effective in the treatment of extensive-stage SCLC after sandard first-line chemotherapy and radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Sign written informed consent;
* With extensive small cell lung cancer;
* Previously received first-line standard chemotherapy, with treatment response of CR or PR;
* Can provide at least 5-8 pathological tissue specimens (for detecting PD-L1 expression and infiltrating lymphocytes)
* Can tolerate the radiotherapy process;
* Weight ≥ 40kg;
* Life expectancy ≥ 12 weeks;
* With the Eastern Cancer Cooperative Group (ECOG) score 0-1;
* The interval from the previous chemotherapy is more than 4 weeks, the grade of all adverse events caused by previous treatment have been reduced to grade 1 or less evaluated by CTCAE 4.03;
* Before the administration of the study drug, systemic drugs (such as corticosteroids) applied at an immunosuppressive dose level (prednisone > 10 mg/d or equivalent) must have been discontinued for at least 2 weeks;
* Major surgery requiring general anesthesia must have been completed for at least 4 weeks before administration of the study drug. Surgery requiring local anesthesia/epidural anesthesia must have been completed for at least 72 hours before administration of the study drug, and the subject must have recovered. Skin biopsy with only local anesthesia has been completed for at least 1 hour before administration of the study drug.
* Other criteria including the laboratory values meets the requirements specified in the protocol.

Exclusion Criteria:

* Subjects with central nervous system (CNS) metastases;
* The subject has cancerous meningitis;
* Subjects with active, known or suspected autoimmune diseases ;
* Previously treated with anti-PD-1 antibody, anti-PD-L1 antibody, anti-PD-L2 antibody or anti-CTLA-4 antibody (or any other antibody acting on the T cell stimulation or checkpoint pathway);
* According to chest X-ray examination, sputum examination and clinical examination, it is determined that there is active tuberculosis (TB) infection now or before, even one year before;
* A positive immunodeficiency virus (HIV) test or have acquired immunodeficiency syndrome (AIDS);
* With comorbidity needs to be treated with an immunosuppressive drug;
* Other research drugs were administrated 28 days prior to the start of study drug or although they were more than 28 days apart, still within the 5 half-life of previous study drugs;
* Inoculated with any anti-infective vaccine (such as influenza vaccine, varicella vaccine, etc.) within 4 weeks before starting the study drug;
* In the condition of pregnant or breastfeeding;
* Inability to tolerate venous puncture and/or venous access;
* Any other medical, psychotic, and/or social problems determined by the investigator;
* Subject has interstitial lung disease;
* Use any Chinese medicine with anti-tumor activity within 2 weeks before starting of the study drug;
* Monoclonal antibodies have been used in the past 3 months, except for topical use;
* Subjects who have previously had other malignancies (excluding non-melanoma skin cancer and the following carcinomas in situ: bladder, stomach, colon, endometrium, cervix/dysplasia, melanoma or breast cancer) are not allowed to participate in the study. Unless he/she has been cured at least 2 years prior to enrollment, and does not require additional treatment or other treatments during the study;
* Subjects with chronic hepatitis B (hepatitis B surface antigen positive) or chronic hepatitis C (HCV antibody positive) blood screening positive;
* Previously allergic to macromolecular protein preparations, or to any of the JS001 ingredients.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2019-06 (Estimated); Primary Completion 2020-06 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Adverse events | At least 1 year following the conclusion of immunotherapy
  The incidence and severity of adverse events related to treatments
Objective remission rate | 24 weeks following the conclusion of immunotherapy
  Objective remission rate (ORR): refers to the proportion of subjects in the analyzed population who achieved complete remission (CR) or partial remission (PR); according to the tumor immunotherapy efficacy evaluation (irRC) and RECIST criteria (v1.1) by the evaluation of investigator.

SECONDARY OUTCOMES:
Pharmacodynamic indicators | During and 6 weeks after the treatment of immunotherapy
  Pharmacodynamic indicators，such as the detection of PD-1 receptor occupancy in the blood
Continuous remission time (DOR) | At least 1 year following the conclusion of immunotherapy
  DOR was defined as time since onset of CR or PR to relapse or death due to underlying cancer, whichever is earlier
Disease Control Rate (DCR) | At least 1 year following the conclusion of immunotherapy
  The percentage of patients who have achieved complete response, partial response and stable disease to the therapeutic intervention
Time to response (TTR) | 24 weeks following the conclusion of immunotherapy
  The time from the start of treatment to the first objective tumor response
Progression-free survival (PFS) | At least 1 year following the conclusion of immunotherapy
  The length of time during and after the treatment of a disease that a patient lives with the disease but it does not get worse
Overall survival (OS) | At least 1 year following the conclusion of immunotherapy
  The time from treatment to death from any cause

OTHER OUTCOMES:
Exploratory end point including biomarkers | At least 1 year following the conclusion of immunotherapy
  To explore the correlation of PD-L1 expression in tumor tissue , TCR, ctDNA in peripheral blood and efficacy

CONTACTS AND LOCATIONS:
Overall Officials: Nan Bi, MD, Study Director — Cancer Hospital, CAMS and PUMC
Locations (1):
- Cancer Insititute and Hosiptal of Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Torre LA, Bray F, Siegel RL, Ferlay J, Lortet-Tieulent J, Jemal A. Global cancer statistics, 2012. CA Cancer J Clin. 2015 Mar;65(2):87-108. doi: 10.3322/caac.21262. Epub 2015 Feb 4. PMID 25651787
- [Background] Chen W, Zheng R, Zhang S, Zeng H, Zuo T, Xia C, Yang Z, He J. Cancer incidence and mortality in China in 2013: an analysis based on urbanization level. Chin J Cancer Res. 2017 Feb;29(1):1-10. doi: 10.21147/j.issn.1000-9604.2017.01.01. PMID 28373748
- [Background] Takada M, Fukuoka M, Kawahara M, Sugiura T, Yokoyama A, Yokota S, Nishiwaki Y, Watanabe K, Noda K, Tamura T, Fukuda H, Saijo N. Phase III study of concurrent versus sequential thoracic radiotherapy in combination with cisplatin and etoposide for limited-stage small-cell lung cancer: results of the Japan Clinical Oncology Group Study 9104. J Clin Oncol. 2002 Jul 15;20(14):3054-60. doi: 10.1200/JCO.2002.12.071. PMID 12118018
- [Background] Turrisi AT 3rd, Kim K, Blum R, Sause WT, Livingston RB, Komaki R, Wagner H, Aisner S, Johnson DH. Twice-daily compared with once-daily thoracic radiotherapy in limited small-cell lung cancer treated concurrently with cisplatin and etoposide. N Engl J Med. 1999 Jan 28;340(4):265-71. doi: 10.1056/NEJM199901283400403. PMID 9920950
- [Background] Janne PA, Freidlin B, Saxman S, Johnson DH, Livingston RB, Shepherd FA, Johnson BE. Twenty-five years of clinical research for patients with limited-stage small cell lung carcinoma in North America. Cancer. 2002 Oct 1;95(7):1528-38. doi: 10.1002/cncr.10841. PMID 12237922
- [Background] Govindan R, Page N, Morgensztern D, Read W, Tierney R, Vlahiotis A, Spitznagel EL, Piccirillo J. Changing epidemiology of small-cell lung cancer in the United States over the last 30 years: analysis of the surveillance, epidemiologic, and end results database. J Clin Oncol. 2006 Oct 1;24(28):4539-44. doi: 10.1200/JCO.2005.04.4859. PMID 17008692
- [Background] Socinski MA, Smit EF, Lorigan P, Konduri K, Reck M, Szczesna A, Blakely J, Serwatowski P, Karaseva NA, Ciuleanu T, Jassem J, Dediu M, Hong S, Visseren-Grul C, Hanauske AR, Obasaju CK, Guba SC, Thatcher N. Phase III study of pemetrexed plus carboplatin compared with etoposide plus carboplatin in chemotherapy-naive patients with extensive-stage small-cell lung cancer. J Clin Oncol. 2009 Oct 1;27(28):4787-92. doi: 10.1200/JCO.2009.23.1548. Epub 2009 Aug 31. PMID 19720897
- [Background] Lara PN Jr, Natale R, Crowley J, Lenz HJ, Redman MW, Carleton JE, Jett J, Langer CJ, Kuebler JP, Dakhil SR, Chansky K, Gandara DR. Phase III trial of irinotecan/cisplatin compared with etoposide/cisplatin in extensive-stage small-cell lung cancer: clinical and pharmacogenomic results from SWOG S0124. J Clin Oncol. 2009 May 20;27(15):2530-5. doi: 10.1200/JCO.2008.20.1061. Epub 2009 Apr 6. PMID 19349543
- [Background] Rossi A, Di Maio M, Chiodini P, Rudd RM, Okamoto H, Skarlos DV, Fruh M, Qian W, Tamura T, Samantas E, Shibata T, Perrone F, Gallo C, Gridelli C, Martelli O, Lee SM. Carboplatin- or cisplatin-based chemotherapy in first-line treatment of small-cell lung cancer: the COCIS meta-analysis of individual patient data. J Clin Oncol. 2012 May 10;30(14):1692-8. doi: 10.1200/JCO.2011.40.4905. Epub 2012 Apr 2. PMID 22473169
- [Background] Slotman BJ, van Tinteren H, Praag JO, Knegjens JL, El Sharouni SY, Hatton M, Keijser A, Faivre-Finn C, Senan S. Use of thoracic radiotherapy for extensive stage small-cell lung cancer: a phase 3 randomised controlled trial. Lancet. 2015 Jan 3;385(9962):36-42. doi: 10.1016/S0140-6736(14)61085-0. Epub 2014 Sep 14. PMID 25230595
- [Background] Slotman BJ, van Tinteren H, Praag JO, Knegjens JL, El Sharouni SY, Hatton M, Keijser A, Faivre-Finn C, Senan S. Radiotherapy for extensive stage small-cell lung cancer - Authors' reply. Lancet. 2015 Apr 4;385(9975):1292-3. doi: 10.1016/S0140-6736(15)60679-1. No abstract available. PMID 25890910
- [Background] Pardoll DM. The blockade of immune checkpoints in cancer immunotherapy. Nat Rev Cancer. 2012 Mar 22;12(4):252-64. doi: 10.1038/nrc3239. PMID 22437870
- [Background] Keir ME, Butte MJ, Freeman GJ, Sharpe AH. PD-1 and its ligands in tolerance and immunity. Annu Rev Immunol. 2008;26:677-704. doi: 10.1146/annurev.immunol.26.021607.090331. PMID 18173375
- [Background] Nishimura H, Agata Y, Kawasaki A, Sato M, Imamura S, Minato N, Yagita H, Nakano T, Honjo T. Developmentally regulated expression of the PD-1 protein on the surface of double-negative (CD4-CD8-) thymocytes. Int Immunol. 1996 May;8(5):773-80. doi: 10.1093/intimm/8.5.773. PMID 8671666
- [Background] Taube JM, Anders RA, Young GD, Xu H, Sharma R, McMiller TL, Chen S, Klein AP, Pardoll DM, Topalian SL, Chen L. Colocalization of inflammatory response with B7-h1 expression in human melanocytic lesions supports an adaptive resistance mechanism of immune escape. Sci Transl Med. 2012 Mar 28;4(127):127ra37. doi: 10.1126/scitranslmed.3003689. PMID 22461641
- [Background] Iwai Y, Ishida M, Tanaka Y, Okazaki T, Honjo T, Minato N. Involvement of PD-L1 on tumor cells in the escape from host immune system and tumor immunotherapy by PD-L1 blockade. Proc Natl Acad Sci U S A. 2002 Sep 17;99(19):12293-7. doi: 10.1073/pnas.192461099. Epub 2002 Sep 6. PMID 12218188
- [Background] Borghaei H, Paz-Ares L, Horn L, Spigel DR, Steins M, Ready NE, Chow LQ, Vokes EE, Felip E, Holgado E, Barlesi F, Kohlhaufl M, Arrieta O, Burgio MA, Fayette J, Lena H, Poddubskaya E, Gerber DE, Gettinger SN, Rudin CM, Rizvi N, Crino L, Blumenschein GR Jr, Antonia SJ, Dorange C, Harbison CT, Graf Finckenstein F, Brahmer JR. Nivolumab versus Docetaxel in Advanced Nonsquamous Non-Small-Cell Lung Cancer. N Engl J Med. 2015 Oct 22;373(17):1627-39. doi: 10.1056/NEJMoa1507643. Epub 2015 Sep 27. PMID 26412456
- [Background] Robert C, Schachter J, Long GV, Arance A, Grob JJ, Mortier L, Daud A, Carlino MS, McNeil C, Lotem M, Larkin J, Lorigan P, Neyns B, Blank CU, Hamid O, Mateus C, Shapira-Frommer R, Kosh M, Zhou H, Ibrahim N, Ebbinghaus S, Ribas A; KEYNOTE-006 investigators. Pembrolizumab versus Ipilimumab in Advanced Melanoma. N Engl J Med. 2015 Jun 25;372(26):2521-32. doi: 10.1056/NEJMoa1503093. Epub 2015 Apr 19. PMID 25891173
- [Background] Antonia SJ, Lopez-Martin JA, Bendell J, Ott PA, Taylor M, Eder JP, Jager D, Pietanza MC, Le DT, de Braud F, Morse MA, Ascierto PA, Horn L, Amin A, Pillai RN, Evans J, Chau I, Bono P, Atmaca A, Sharma P, Harbison CT, Lin CS, Christensen O, Calvo E. Nivolumab alone and nivolumab plus ipilimumab in recurrent small-cell lung cancer (CheckMate 032): a multicentre, open-label, phase 1/2 trial. Lancet Oncol. 2016 Jul;17(7):883-895. doi: 10.1016/S1470-2045(16)30098-5. Epub 2016 Jun 4. PMID 27269741
- [Background] Stone HB, Peters LJ, Milas L. Effect of host immune capability on radiocurability and subsequent transplantability of a murine fibrosarcoma. J Natl Cancer Inst. 1979 Nov;63(5):1229-35. No abstract available. PMID 291749
- [Background] Formenti SC, Demaria S. Combining radiotherapy and cancer immunotherapy: a paradigm shift. J Natl Cancer Inst. 2013 Feb 20;105(4):256-65. doi: 10.1093/jnci/djs629. Epub 2013 Jan 4. PMID 23291374
- [Background] Sharabi AB, Lim M, DeWeese TL, Drake CG. Radiation and checkpoint blockade immunotherapy: radiosensitisation and potential mechanisms of synergy. Lancet Oncol. 2015 Oct;16(13):e498-509. doi: 10.1016/S1470-2045(15)00007-8. PMID 26433823
- [Background] Dovedi SJ, Adlard AL, Lipowska-Bhalla G, McKenna C, Jones S, Cheadle EJ, Stratford IJ, Poon E, Morrow M, Stewart R, Jones H, Wilkinson RW, Honeychurch J, Illidge TM. Acquired resistance to fractionated radiotherapy can be overcome by concurrent PD-L1 blockade. Cancer Res. 2014 Oct 1;74(19):5458-68. doi: 10.1158/0008-5472.CAN-14-1258. PMID 25274032
- [Background] Deng L, Liang H, Burnette B, Beckett M, Darga T, Weichselbaum RR, Fu YX. Irradiation and anti-PD-L1 treatment synergistically promote antitumor immunity in mice. J Clin Invest. 2014 Feb;124(2):687-95. doi: 10.1172/JCI67313. Epub 2014 Jan 2. PMID 24382348
- [Background] Sharabi AB, Nirschl CJ, Kochel CM, Nirschl TR, Francica BJ, Velarde E, Deweese TL, Drake CG. Stereotactic Radiation Therapy Augments Antigen-Specific PD-1-Mediated Antitumor Immune Responses via Cross-Presentation of Tumor Antigen. Cancer Immunol Res. 2015 Apr;3(4):345-55. doi: 10.1158/2326-6066.CIR-14-0196. Epub 2014 Dec 19. PMID 25527358
- [Background] Verbrugge I, Hagekyriakou J, Sharp LL, Galli M, West A, McLaughlin NM, Duret H, Yagita H, Johnstone RW, Smyth MJ, Haynes NM. Radiotherapy increases the permissiveness of established mammary tumors to rejection by immunomodulatory antibodies. Cancer Res. 2012 Jul 1;72(13):3163-74. doi: 10.1158/0008-5472.CAN-12-0210. Epub 2012 May 8. PMID 22570253
- [Background] Zeng J, See AP, Phallen J, Jackson CM, Belcaid Z, Ruzevick J, Durham N, Meyer C, Harris TJ, Albesiano E, Pradilla G, Ford E, Wong J, Hammers HJ, Mathios D, Tyler B, Brem H, Tran PT, Pardoll D, Drake CG, Lim M. Anti-PD-1 blockade and stereotactic radiation produce long-term survival in mice with intracranial gliomas. Int J Radiat Oncol Biol Phys. 2013 Jun 1;86(2):343-9. doi: 10.1016/j.ijrobp.2012.12.025. Epub 2013 Feb 22. PMID 23462419
- [Background] Ahmed KA, Stallworth DG, Kim Y, Johnstone PA, Harrison LB, Caudell JJ, Yu HH, Etame AB, Weber JS, Gibney GT. Clinical outcomes of melanoma brain metastases treated with stereotactic radiation and anti-PD-1 therapy. Ann Oncol. 2016 Mar;27(3):434-41. doi: 10.1093/annonc/mdv622. Epub 2015 Dec 27. PMID 26712903
- [Background] Shaverdian N, Lisberg AE, Bornazyan K, Veruttipong D, Goldman JW, Formenti SC, Garon EB, Lee P. Previous radiotherapy and the clinical activity and toxicity of pembrolizumab in the treatment of non-small-cell lung cancer: a secondary analysis of the KEYNOTE-001 phase 1 trial. Lancet Oncol. 2017 Jul;18(7):895-903. doi: 10.1016/S1470-2045(17)30380-7. Epub 2017 May 24. PMID 28551359
- [Background] Antonia SJ, Villegas A, Daniel D, Vicente D, Murakami S, Hui R, Yokoi T, Chiappori A, Lee KH, de Wit M, Cho BC, Bourhaba M, Quantin X, Tokito T, Mekhail T, Planchard D, Kim YC, Karapetis CS, Hiret S, Ostoros G, Kubota K, Gray JE, Paz-Ares L, de Castro Carpeno J, Wadsworth C, Melillo G, Jiang H, Huang Y, Dennis PA, Ozguroglu M; PACIFIC Investigators. Durvalumab after Chemoradiotherapy in Stage III Non-Small-Cell Lung Cancer. N Engl J Med. 2017 Nov 16;377(20):1919-1929. doi: 10.1056/NEJMoa1709937. Epub 2017 Sep 8. PMID 28885881
- [Background] Schaue D, Ratikan JA, Iwamoto KS, McBride WH. Maximizing tumor immunity with fractionated radiation. Int J Radiat Oncol Biol Phys. 2012 Jul 15;83(4):1306-10. doi: 10.1016/j.ijrobp.2011.09.049. Epub 2011 Dec 28. PMID 22208977
- [Background] Dewan MZ, Galloway AE, Kawashima N, Dewyngaert JK, Babb JS, Formenti SC, Demaria S. Fractionated but not single-dose radiotherapy induces an immune-mediated abscopal effect when combined with anti-CTLA-4 antibody. Clin Cancer Res. 2009 Sep 1;15(17):5379-88. doi: 10.1158/1078-0432.CCR-09-0265. Epub 2009 Aug 25. PMID 19706802
- [Background] Finkelstein SE, Timmerman R, McBride WH, Schaue D, Hoffe SE, Mantz CA, Wilson GD. The confluence of stereotactic ablative radiotherapy and tumor immunology. Clin Dev Immunol. 2011;2011:439752. doi: 10.1155/2011/439752. Epub 2011 Nov 15. PMID 22162711